CLINICAL TRIAL: NCT04051814
Title: A Retrospective Trial to Evaluate the Micra Pacemaker
Acronym: Micra
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Principal Investigator, Colleen Balius, Clinical Data Coordinator, Hoag Memorial Hospital Presbyterian
Other Study IDs: 191-18-CV
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Pacemaker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Micra Transcatheter Pacemaker System — A miniaturized single chamber pacemaker system that is delivered via catheter through the femoral vein and is implanted directly inside the right ventricle of the heart

SUMMARY:
This is a retrospective study of our patient population implanted with the Medtronic's Leadless single-chamber ventricular pacemakers.

DETAILED DESCRIPTION:
This protocol outlines the methods on the Micra Pacemaker. The Micra Transcatheter Pacemaker System is a miniaturized single chamber pacemaker system that is delivered via catheter through the femoral vein and is implanted directly inside the right ventricle of the heart. The Micra device eliminates the need for a device pocket and insertion of a pacing lead, thereby eliminating lead and pocket related complications associated with traditional pacing systems while providing similar pacing benefits. The US Food and Drug Administration (FDA) approved the Micra system on April 6, 2016, for the following conditions:

* symptomatic paroxysmal or permanent high-grade atrioventricular block (AV) in the presence of atrial fibrillation (AF)
* symptomatic paroxysmal or permanent high-grade AV block in the absence of AF, as an alternative to dual chamber pacing, when atrial lead placement is considered difficult, high risk, or not deemed necessary for effective therapy
* symptomatic bradycardia-tachycardia syndrome or sinus node dysfunction (sinus bradycardia or sinus pauses), as an alternative to atrial or dual chamber pacing, when atrial lead placement is considered difficult, high risk, or not deemed necessary for effective therapy The FDA approved the Micra system on the basis of clinical trial evidence from the Micra Investigational Device Exemption (IDE) study (NCT02488681).

On January 18, 2017, the Centers for Medicare and Medicaid Services (CMS) issued a final National Coverage Determination (NCD) on leadless pacemakers, providing for coverage with Coverage with Evidence Development (CED) of approved leadless pacemakers for approved indications (CAG-00448N). The NCD requires the research study conducted as part of CED to address the following research questions:

1. What are the peri-procedural and post-procedural complications of leadless pacemakers?
2. What are the long-term outcomes of leadless pacemakers?
3. What are the effects of patient characteristics (age, gender, comorbidities) on the use and health effects of leadless pacemakers?

In addition, CMS outlined six evidentiary gaps in the final NCD for leadless pacemakers:

1. What are the peri-procedural and post-procedural complications, and long term outcomes of leadless pacemakers?
2. Are leadless pacemakers equivalent or superior to conventional pacemaker's in general clinical practice?
3. What are the infection rates, the long-term hemodynamic effects, and the rates of formation of thrombi?
4. What are the patient demographics and effects of patient characteristics (age, gender, comorbidities) on the use and health effects of leadless pacemakers?
5. What are the device-related issues (handling of end of battery life; effects of having multiple leadless pacemakers implanted; rate of device dislodgement; and the possibility of device extractions)?
6. How are operators and facility characteristics related to peri-procedural and post-procedural complications?

ELIGIBILITY:
Inclusion Criteria:

* All Patients scheduled to be implanted with a leadless pacemaker

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Patients scheduled to be implanted with a leadless pacemaker
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-07-31 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Complication Rate | 2 years
  We plan to collect data to determine the acute overall complication rate

CONTACTS AND LOCATIONS:
Locations (1):
- Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: Undecided